CLINICAL TRIAL: NCT04774705
Title: Randomized Pilot Study Evaluating the Effectiveness of Non-invasive Vagus Nerve Stimulation as an Adjuvant Treatment in Patients With Sepsis in Intensive Care.
Brief Title: Effectiveness of Non-invasive Vagus Nerve Stimulation as an Adjuvant Treatment in Patients With Sepsis in Intensive Care.
Acronym: SNV-Sepsis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: D20170804
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNV activ group (Non-invasive transcutaneous stimulation of the vagus nerve ) (Experimental)
  Interventions: Other: SNV activ group (Non-invasive transcutaneous stimulation of the vagus nerve )
- Control group (Placebo Comparator): For the SNV placebo group, the stimulation electrode will be inverted so as to deliver the stimulation to the ear lobule.
  Interventions: Other: Placebo group

INTERVENTIONS:
Other: SNV activ group (Non-invasive transcutaneous stimulation of the vagus nerve ) — A transcutaneous stimulator of the atrial branch of the vagus nerve of the TENS eco Plus type (Schwa-medico) will be used. SNV stimulation will be applied in the concha of the left ear to the subcutaneous area of the atrial branch of the vagus nerve in the left ear (cymba conchae) for each patient, at an intensity of 2 mA, 30 minutes per day for 5 consecutive days, from the day of inclusion / randomization.
  Arms: SNV activ group (Non-invasive transcutaneous stimulation of the vagus nerve )
Other: Placebo group — For the control group, the stimulation electrode will be inverted so as to deliver the stimulation to the ear lobule.
  Arms: Control group

SUMMARY:
Sepsis is one of the leading causes of death in intensive care. About 50% of patients with septic shock die after 1 year; and 50% of survivors suffer from cognitive decline. The pathophysiological mechanisms of serious complications of sepsis are now well known. In fact, the systemic inflammation related to sepsis amplifies the release of pro-inflammatory cytokines and neurotoxic mediators, hence an increase in deleterious phenomena such as oxidative stress, mitochondrial dysfunction, endothelial activation, disruption of the blood-brain barrier, neuroinflammation (astrocytic and microglial activation) leading to multi-organ failure which compromises the patient's vital and functional prognosis. Although there has been progress in the understanding of its pathophysiology, the management of sepsis and septic shock in intensive care relies mainly on anti-infective treatments and the restoration of cardiovascular and respiratory functions. There is virtually no adjuvant therapy for the management of sepsis, apart from a few hormonal therapies such as insulin to maintain blood glucose levels below 180 mg / dL and low doses of corticosteroids and vasopressin. There is therefore a pressing need to develop innovative treatments targeting inflammatory and immunological processes in order to reduce the complications of sepsis and improve patient prognosis. Some recent work has shown that electrical vagus nerve stimulation (SNV), a technique used for the treatment of drug-resistant epilepsy, can modulate inflammatory and immune responses and control inflammation syndrome in animal models of sepsis, arthritis and rheumatism in humans. In this pilot study the investigators plan to evaluate the efficacy of transcutaneous (non-invasive) SNV as an adjuvant treatment in patients with sepsis in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years old
* Adult man or woman, hospitalized in intensive care, presenting with sepsis for at least 24 hours according to the diagnostic criteria (Singer et al., 2016).
* Informed consent signed by patient or family member/trusted support person
* In an emergency situation, in the absence of family members/trusted family/trusted support person

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient in a severe state of agitation.
* Patient in a state of brain death or active limitation of treatment.
* Multiple trauma patient, with multiple fractures of the skull.
* Refusal to participate in the study or to sign the informed consent by the patient or his loved one,
* Pregnant or breastfeeding woman,
* No affiliation to a social security scheme.
* Patient with cochlear implant
* Patient with heart disease
* Patient with asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2025-03-29 (Estimated); Study Completion 2025-03-29 (Estimated)

PRIMARY OUTCOMES:
Mortality | at day 90
  Overall death

SECONDARY OUTCOMES:
Cumulative incidence of delirium and its duration | up to day 90
Cumulative incidence of mechanical ventilation and its duration | up to day 90
Proportion of patients having been the subject of a decision to limit or withdraw care | at day 90
Duration of use of vasopressors | at day 90
Number of days alive with a Sequential Organ Failure Assessment Score (SOFA) score <6 | at day 90
  Sequential Organ Failure Assessment Score varies from 0 to 4 and permit to assess organ failure. A higher score indicates better neurological function
Length of stay in intensive care and hospitalization in all patients and in survivors | at day 90
Measurements of changes in C-reactive protein (CRP) | at inclusion
Measurements of changes in C-reactive protein (CRP) | at day 7
Measurements of changes in C-reactive protein (CRP) | at day 14
Measurements of changes in C-reactive protein (CRP) | at day 21
Measurements of changes in C-reactive protein (CRP) | at day 28
Measurements of changes in C-reactive protein (CRP) | at day 90
Measurements of changes in fibrinogen level | at inclusion
Measurements of changes in fibrinogen level | at day 7
Measurements of changes in fibrinogen level | at day 14
Measurements of changes in fibrinogen level | at day 21
Measurements of changes in fibrinogen level | at day 28
Measurements of changes in fibrinogen level | at day 90
Measurements of changes in interleukin-6 (IL-6) | at inclusion
Measurements of changes in interleukin-6 (IL-6) | at day 7
Measurements of changes in interleukin-6 (IL-6) | at day 14
Measurements of changes in interleukin-6 (IL-6) | at day 21
Measurements of changes in interleukin-6 (IL-6) | at day 28
Measurements of changes in interleukin-6 (IL-6) | at day 90
Measurements of changes in interleukin-1β (IL-1β) | at inclusion
Measurements of changes in interleukin-1β (IL-1β) | at day 7
Measurements of changes in interleukin-1β (IL-1β) | at day 14
Measurements of changes in interleukin-1β (IL-1β) | at day 21
Measurements of changes in interleukin-1β (IL-1β) | at day 28
Measurements of changes in interleukin-1β (IL-1β) | at day 90
Measurements of changes in tumor necrosis factor α (TNF-α) | at inclusion
Measurements of changes in tumor necrosis factor α (TNF-α) | at day 7
Measurements of changes in tumor necrosis factor α (TNF-α) | at day 14
Measurements of changes in tumor necrosis factor α (TNF-α) | at day 21
Measurements of changes in tumor necrosis factor α (TNF-α) | at day 28
Measurements of changes in tumor necrosis factor α (TNF-α) | at day 90
Measurements of changes in the calcium binding protein B S100B (S100B) | at inclusion
Measurements of changes in the calcium binding protein B S100B (S100B) | at day 7
Measurements of changes in the calcium binding protein B S100B (S100B) | at day 14
Measurements of changes in the calcium binding protein B S100B (S100B) | at day 21
Measurements of changes in the calcium binding protein B S100B (S100B) | at day 28
Measurements of changes in the calcium binding protein B S100B (S100B) | at day 90
Measurements of changes in the arterial lactate level | at inclusion
Measurements of changes in the arterial lactate level | at day 7
Measurements of changes in the arterial lactate level | at day 14
Measurements of changes in the arterial lactate level | at day 21
Measurements of changes in the arterial lactate level | at day 28
Measurements of changes in the arterial lactate level | at day 90
Characteristics of the EEG | at inclusion
Characteristics of the EEG | at day 7
Mortality rate | at day 28
  Overall death
Neurological fate of patients | at day 90
  Neurological fate of patients will evaluated using Glasgow Outcome Scale (GOS)

CONTACTS AND LOCATIONS:
Locations (1):
- Raymond Poincaré Hospital, Garches, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goggins E, Inoue H, Okusa MD. Neuroimmune Control of Inflammation in Acute Kidney Injury and Multiorgan Dysfunction. J Am Soc Nephrol. 2025 Dec 1;36(12):2473-2484. doi: 10.1681/ASN.0000000813. Epub 2025 Jul 7. PMID 40622772